CLINICAL TRIAL: NCT03740074
Title: Evaluation of Personal Activity Intelligence (PAI) Score Pilot Study
Brief Title: Personal Activity Intelligence (PAI) Pilot
Acronym: PAI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio University (Other)
Responsible Party: Principal Investigator, David Drozek, Associate Professor, Ohio University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-X-263
Record Dates: First submitted 2018-11-08; First posted 2018-11-14 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Overweight and Obesity; Diabetes; Hypertension; Dyslipidemias; Cardiovascular Diseases
MeSH Terms: conditions — Overweight; Obesity; Diabetes Mellitus; Hypertension; Dyslipidemias; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Prospective pilot
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PAI (Experimental): Participants will utilize a MIO Slice wearable device to generate a PAI score, which will be utilized to provide feedback and incentive for physical activity.
  Interventions: Behavioral: PAI

INTERVENTIONS:
Behavioral: PAI — Consenting subjects will be given a Mio Slice, along with instructions on how to utilize the device.
  They will register on line with PAI Health, and will be asked to sync their device at least once every 7 days. They will be encouraged to look at the device app on their smart phone at least once daily.
  After 1 week of obtaining baseline data, subjects will be encouraged to try to obtain a PAI score of at least 30 initially. Once they obtain a score of 30 consistently, they will be encouraged to increase the score toward 50. If they consistently obtain 50, they can increase their goal sequentially toward a maximum goal of 100. The duration of the study will be 12 weeks.

SUMMARY:
Pilot study to evaluate the use of the Personal Activity Intelligence (PAI) score in a clinical setting.

DETAILED DESCRIPTION:
This is a pilot project to evaluate the feasibility of a larger study to evaluate the effectiveness of Personal Activity Intelligence (PAI) score in patients with chronic disease, as an adjunct to lifestyle medical therapy.

The PAI score is a proprietary formula developed by PAI Health (PH) to aid physical fitness. A PAI score calculation uses biometrics obtained via a device that measures heart rate and steps. For this study, Mio Slice, a commercial wrist worn device will be utilized to obtain data which will be linked to a smart phone. Data from the smart phone app will be accessed by PAI Health. Feedback information will be given to the participants to encourage increased physical activity.

The short-term aim of this study is to evaluate the logistics of utilizing PAI in the patient setting.

The data obtained from this study will be utilized to devise a larger study to evaluate the utility of PAI in patients with chronic disease who are receiving lifestyle medical therapy.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who are seen by the PI in his lifestyle medicine practice at Muntean Health Care.
* Participants must own a smart phone and feel comfortable managing apps on their smart phone.
* Participants must be willing and able to register online with PAI Health (PH)
* Participants must be willing to wear a wrist device around the clock, except when charging or bathing for 12 weeks.
* Participants must have at least one of the following diagnoses:
* overweight / obesity
* diabetes or prediabetes
* hypertension or pre-hypertension
* abnormal lipids
* cardiovascular disease

Exclusion Criteria:

* Patients with angina or poor exercise tolerance, based on the evaluation by the PI, will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-10-02 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
App utility | 12 weeks
  ease in use of obtaining and using PAI score by the patient based on a patient survey

SECONDARY OUTCOMES:
Systolic blood pressure | 12 weeks
  change in systolic blood pressure
Diastolic blood pressure | 12 weeks
  change in diastolic blood pressure
Weight | 12 weeks
  change in weight
Personal Activity Intelligence (PAI) Score | 12 weeks
  The Personal Activity Intelligence (PAI) Score is a proprietary calculation owned by PAI Health, and not made available to the investigator. The score does take in to account resting heart rate while sleeping, peak heart rate during physical activity, length of time of elevated heart rate, steps. This data is captured via a wearable device, Mio Slice which is synced with a smart phone. Participants are encouraged to keep their PAI Score at 100, or as high as possible.

CONTACTS AND LOCATIONS:
Overall Officials: David S Drozek, DO, Principal Investigator — Ohio University
Locations (1):
- Ohio University, Athens, Ohio, United States